CLINICAL TRIAL: NCT02226328
Title: Nurse Administered Propofol Sedation vs. Midazolam With Fentanyl-sedation for Flexible Bronchoscopy: A Randomized, Single Blind, Controlled Study of Satisfaction and Safety.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-004358-12
Record Dates: First submitted 2014-08-19; First posted 2014-08-27 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Flexible Bronchoscopy; Sedation; Satisfaction; Safety
MeSH Terms: conditions — Personal Satisfaction | interventions — Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol sedation (Experimental): Refract bolus propofol sedation as monotherapy administered by a sedation-trained nurse endoscopist.
  Induction with 10-60 mg bolus, repeated every 45-60 sec. until moderate sedation.
  Maintenance with 10-20 mg of propofol in case of discomfort.
  Interventions: Drug: Propofol sedation
- Midazolam and Fentanyl sedation (Active Comparator): 1-2 mg of Midazolam with 0.025-0.05 mg of fentanyl for induction 10 prior to procedure initiation.
  Maintenance with 1 mg Midazolam in case of discomfort.
  Interventions: Drug: Midazolam and Fentanyl sedation

INTERVENTIONS:
Drug: Propofol sedation
  Other Names: ATC code: N01AX10; CAS no: 2078-54-8
  Arms: Propofol sedation
Drug: Midazolam and Fentanyl sedation
  Other Names: Midazolam:; ATC code: N05CD08; CAS no: 59467-70-8; Fentanyl:; ATC code: N01AH01; CAS no: 437-38-7
  Arms: Midazolam and Fentanyl sedation

SUMMARY:
Flexible bronchoscopy almost always requires sedation to be successful. In order to increase the availability of propofol for sedation, non-anaesthesiologist administered propofol sedation has been suggested as an alternative to traditional midazolam/opioid sedation or the general anaesthesia provided by anaesthesiologists.

Hypothesis: Patients undergoing flexible bronchoscopy prefers non-anaesthesiologist administered sedation with propofol as opposed to non-anaesthesiologist administered sedation with midazolam and fentanyl.

Propofol sedation is as safe as midazolam and fentanyl sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Elective flexible bronchoscopy.
2. Willing to be randomised
3. Provide written informed consent

Exclusion Criteria:

1. Allergy to contents administered
2. pregnant or nursing
3. <18 years of age
4. Not able to complete questionnaire
5. Acute condition
6. severe COPD
7. > ASA II
8. Sleep apnea
9. Risk of aspiration
10. Previously difficulty with anesthesia
11. Difficult airway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with sedation | At discharge, on average 30 minutes after procedure termination.
  The average duration of bronchoscopy is estimated to 20 minutes. A validated satisfaction questionnaire will be filled by the patient at discharge from the recovery room, on average 30 minutes after completed procedure. Readiness for discharge will be assessed using an Aldrete score.

SECONDARY OUTCOMES:
Number of adverse events as a surrogate marker of safety. | During procedure. On average 20 minutes.
  Adverse events as a dichotomous value of "no event" or "event". Events are: The use of rescue medicine, and cardiopulmonary support per-operatively, blood pressure deviation from baseline over 30% of Mean Arterial Pressure, oxygen saturation < 90%, and arrhythmias will be recorded for the duration of the procedure.

OTHER OUTCOMES:
Patient comfort | Per-operatively, on average 20 minutes
  Patient discomfort/comfort will be registered on a validated scale during the procedure and recorded by the endoscopy nurse. If the procedure was unsuccessful due to discomfort, this will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Clementsen, Professor, Principal Investigator — University of Copenhagen at Gentofte Hospital
Locations (1):
- Gentofte Hospital, Hellerup, Denmark